CLINICAL TRIAL: NCT05888285
Title: Is Radiofrequency Necessary in Myofascial Pain?
Brief Title: Erector Spina Plane Block and Radiofrequency Treatmen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Director, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ESP Block VS ESP RF
Record Dates: First submitted 2023-05-15; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Back Pain; Block; Pain, Muscle
MeSH Terms: conditions — Back Pain; Bites and Stings; Myalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP Block (Active Comparator): ESP block for back pain treatment is applied
  Interventions: Procedure: Erector spina plane block
- ESP RFT (Active Comparator): ESP block and pulsed radiofrequency for back pain treatment is applied
  Interventions: Procedure: Erector spina bale block and pulsed radiofrequency

INTERVENTIONS:
Procedure: Erector spina plane block — The transverse processes of the thoracic vertebrae are treated with ultrasound-guided drug injection
  Arms: ESP Block
Procedure: Erector spina bale block and pulsed radiofrequency — The transverse processes of the thoracic vertebrae are treated with ultrasound-guided drug injection and pulsed radiofrequency treatment
  Arms: ESP RFT

SUMMARY:
ESP is the deepest back muscle originating from the transverse processes of the vertebrae. Blocks applied to this region are effective for a longer time and in the broader area than those applied to superficial muscles. Recently, pulsed radiofrequency treatments have also been performed in myofascial pain, and successful results have been obtained. The investigators aim to investigate whether there is a difference between these two applications in terms of treatment efficacy.

DETAILED DESCRIPTION:
Trigger point injections and erector spina planus muscle (ESP) blocks are used to treat back pain related to myofascial pain syndrome. ESP is the deepest back muscle originating from the transverse processes of the vertebrae. Blocks applied to this region are effective for a longer time and in the broader area than those applied to superficial muscles. Recently, pulsed radiofrequency treatments have also been performed in myofascial pain, and successful results have been obtained.

Deep and superficial back muscles, transverse processes of the vertebrae, costume, and pleural movement are identified by ultrasonographic examination. The investigators perform the intervention through the transverse processes. The investigators give 20 ccs of fluid (bupivacaine, steroids, saline). The patients to whom The investigators apply pulsed radiofrequency complete the procedure by giving 20 ccs of fluid after the radiofrequency application on the transverse processes and during the procedure, using 10 cm, 21 gauge radiofrequency needles with an active tip of 10 mm. The radiofrequency wave is applied at 2 Hz, ten milliseconds, and 55 volts for 5+5 for 10 minutes.

The investigators aim to investigate whether there is a difference between these two applications in terms of treatment efficacy. For this reason, the Visual Pain Scale of each patient will be recorded before the procedure, the second week after the procedure, and the first month. The Centrality of Pain Scale will be applied to these patients at the controls. The correlation between the results of this scale, which evaluates the emotional and physical state of the patients, and the post-treatment pain scales will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* myofascial pain
* normal thoracic examination

Exclusion Criteria:

* additional cardiac disease
* lung disease
* malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-14 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | Change from Baseline VAS at third months.
  It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.

SECONDARY OUTCOMES:
Centrality of pain Scale | Before treatment
  The Centrality of Pain Scale (COPS) is a 10-item self-report measure designed to assess. Each item is scored on a 5-point Likert scale where 1=strongly disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, and 5=strongly agree. Three items are reverse scored the extent to which pain dominates a patient's life.

CONTACTS AND LOCATIONS:
Locations (1):
- Gevher Rabia Genç Perdecioğlu, Ankara, Umit Province, Turkey (Türkiye)